CLINICAL TRIAL: NCT04443179
Title: Brain Imaging and Infant Development
Brief Title: Brain Imaging in Babies Study
Acronym: BIBS
Status: Recruiting | Type: Observational
Sponsor: King's College London (Other)
Responsible Party: Principal Investigator, Dr Grainne McAlonan, Principal Investigator, King's College London
Other Study IDs: IRAS: 108997, REC 12/LO/2017
Record Dates: First submitted 2020-06-19; First posted 2020-06-23 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Autism Spectrum Disorder; Attention Deficit Hyperactivity Disorder; Neurodevelopmental Conditions; COVID-19
MeSH Terms: conditions — Autism Spectrum Disorder; Attention Deficit Disorder with Hyperactivity; COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Infants a family history of ASD/ADHD
- Infants without a family history of ASD/ADHD

SUMMARY:
The aims of the BIBS Study

The Brain Imaging in Babies study (BIBS) aims to improve understanding of how a baby's brain develops from before birth, up until 3-4 years of age. Working with children from a variety of backgrounds and communities, the investigators use a combination of state-of-the-art diagnostic tools such as MRI scans alongside traditional behavioural assessments to capture the earliest information on infant brain development.

The focus of the BIBS study

MRI scanning is a safe way of producing detailed images using strong magnetic fields and radio waves. It does not use X-ray. Along with learning more about brain development in general, the investigators also try to identify features that may in future help predict whether a child will or will not develop traits of conditions such as Autism Spectrum Disorder (ASD) or Attention Deficit Hyperactivity Disorder (ADHD). Long-term, this may help target useful interventions early on, helping children who are most in need.

Since COVID-19 arrived in the United Kingdom (U.K.) in 2020, the investigators have been given ethical approval to include testing for this infection in the mothers and children participating in the study. This may provide an opportunity to better understand how mother and baby respond to infections. The investigators particularly welcome mothers who have had a positive COVID-19 test during their pregnancy to join the study.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant mothers with and without confirmed COVID-19
* Infants with and without an immediate family history of Autism Spectrum and neurodevelopmental conditions
* Based in England, UK

Exclusion Criteria:

* based on further screening

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Community Sample
Sampling Method: Non-Probability Sample
Enrollment: 790 (Estimated)
Dates: Start 2013-04-05 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Neurodevelopmental Outcomes | 3-4 years of age

CONTACTS AND LOCATIONS:
Locations (1):
- King's College London, London, United Kingdom